CLINICAL TRIAL: NCT06576700
Title: Effect of Procyanidins in the Leaky Gut Repairing Associated with Inflammatory Bowel Disease
Brief Title: Effect of Procyanidins in Leaky Gut Repairing in IBD
Acronym: EcoVitis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Padova (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 5908/AO/24
Record Dates: First submitted 2024-08-26; First posted 2024-08-29 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Ulcerative Colitis in Remission
Keywords: Microbiota; proanthocyanidine; polyphenols

STUDY DESIGN:
Intervention Model Description: This is a pilot,open label, single-treatment trial in which the enrolled subjects will be included in a one-year period, after the written informed consent collection. 25 UC patients in remission phase, both males and females, will be included in a one-year period, after the written informed consent collection. Patients will be treated with the Ecovitis extract. Patients will be asked to take 2 capsules per day, away from meals, for 8 weeks. The therapy undertaken could not be changed nor stopped during the supplement administration.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Active supplement (Experimental): Treatment: the capsules contains Grape Seed Extract GSE-0001- Proanthocyanidins <95%)
  Interventions: Biological: Grape Seed Extracts

INTERVENTIONS:
Biological: Grape Seed Extracts — 2 capsules/day for 8 weeks
  Other Names: EcoVitis

SUMMARY:
The goal of this clinical trial is to learn if the Grape Seed Extract Ecovitis, featuring low monomeric catechins content and a high concentration of oligo-polymeric procyanidins, could modulate the Gut Microbiota composition of Ulcerative Colitis patients during the remission phase. The main questions it aims to answer are:

Does Ecovitis improve the microbiota composition in patients with Ulcerative colitis? Is the intestinal permeability affected? What about the variation in the quality of life?

Participants will:

Take 2 capsules/day of Ecovitis for eight weeks Visit the clinic two times for checkups, serum collection, and Questionaire.

DETAILED DESCRIPTION:
The leaky gut is an alteration of the intestinal epithelium capable of compromising the functionality of the intestinal barrier, permitting the entry of foods or viral/bacterial proteins, and then stimulating the immune system's response. This phenomenon leads to the activation of one or more inflammatory cascades, and it has been associated with the development of various pathologies and associated disorders. The leakage in the leaky gut may be responsible for a huge variety of health issues, ranging from minor (bloating, cramps, fatigue, food allergies, sensitivities, gas, and headaches) to "bigger things": autoimmune conditions, depression, and other mood disorders, diabetes, inflammatory bowel disease (IBD), and multiple sclerosis. Recent studies have shown that procyanidins have a protective effect on the intestinal barrier. Procyanidins, as a kind of dietary flavonoid, have excellent pharmacological properties, such as antioxidant, antibacterial, anti-inflammatory, and anti-tumor properties, so they could be used to treat various diseases, including Alzheimer's disease, diabetes, rheumatoid arthritis, tumors, and obesity. In particular, in vitro studies showed that procyanidins act on tight junctions and, for this reason, they could be able to modify the pathogenic cascade of various gastrointestinal pathologies, including those already mentioned, where the leaky gut plays an important role.

Grape Seed Extracts (GSEs) contain variable amounts of polyphenols and so-called oligomeric proanthocyanidins (PACs). GSEs have been investigated in several health conditions, including cardiovascular disease (CVDs) prevention, chronic venous insufficiency (CVI) management, and type 2 diabetes. Finally, it is known that the Intestinal Microbiota plays a decisive role in the degradation of PACs, but it is unknown which is the effect of PACs on the microbiota itself and its metabolic potential.

In this pilot study, the investigators will evaluate the effect of a new grape seed extract on microbiota modulation and leaky gut reduction in IBD patients.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of UC confirmed by clinical, endoscopic and histopathological evidence. Disease in remission phase confirmed by clinical, endoscopic and histopathological evidence.

  * Age between 18 and 75 years old
  * Ability of subject to participate fully in all aspects of this clinical trial.

Exclusion Criteria:

* ● Patients that have active UC, determined by clinical, endoscopic and histopathological evidences

  * Known diagnosis of CD, indeterminate colitis, ischemic colitis, radiation colitis, diverticular disease associated with colitis or microscopic colitis
  * Positive stool culture for active C. difficile
  * Pregnant women
  * Patients under antibiotic and/or probiotic treatment within 10 days prior to Visit 1.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2024-06-15 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-06-12 (Estimated)

PRIMARY OUTCOMES:
● Evaluation of the gut microbiota composition and variation (microbiota test) | 9 months
  Collection of faecal sample for the assessment of the faecal microbiota composition ribosomal ribonucleic acid ( rRNA16S) The 16S rRNA gene is a bacterial ribosomal gene and a part of the 30S subunit which is used in the identification, characterization, and classification of various bacteria. Samples were normalized, pooled, and run on Illumina MiSeq , in order to evaluate the composition of gut microbiota in terms of bacterial diversity ( alfa and beta) and abundance and any variability associated with the treatment.

SECONDARY OUTCOMES:
● Evaluation of intestinal permeability (Leaky Gut-Zonulin test ) | 10 months
  The serum zonulin( normal value 20-48 ng/ml) test allows for the evaluation of intestinal permeability, as zonulin, a protein produced by intestinal cells, when released, causes an increase in the permeability of tight junctions.
● Evaluation of quality of life IBDQ ( test IBDQ) | 10 months
  The validated IBDQ-32 test, consisting of 32 questions related to the quality of life(QoL) of IBD patients, will be proposed. ( IBDQ <170 bad QoL; IBDQ>/= 170 better QoL)

CONTACTS AND LOCATIONS:
Overall Officials: Edoardo V Savarino, MD, PhD, Principal Investigator — University of Padova
Locations (1):
- Edoardo Vincenzo Savarino, Padua, Padua, Italy